CLINICAL TRIAL: NCT00137631
Title: Evaluation of Many Men, Many Voices, A Group Intervention for STD/HIV Prevention for Black Men Who Have Sex With Men (MSM) in the New York Metropolitan Area by People of Color in Crisis, Brooklyn, NY
Brief Title: Evaluation of Many Men, Many Voices, An STD/HIV Prevention Intervention for Black MSM
Acronym: 3MV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of Rochester (Other)
Responsible Party: Executive Director, People of Color in Crisis, Inc.
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CDC-NCHSTP-CCU224517; U65/CCU224517-01 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Results first posted 2010-05-14 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2010-04

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
Keywords: Adult; HIV Infections / pc [Prevention & Control]; Homosexuality, Male; Humans; Male; Risk-Taking; Safe Sex; Sexual Behavior; HIV
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Homosexuality, Male; Risk-Taking; Safe Sex; Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Many Men, Many Voices (3MV) Intervention (Experimental): Receive 6-session intervention immediately after baseline assessment and randomization
  Interventions: Behavioral: Many Men, Many Voices (3MV)
- Wait list comparison (No Intervention): Receive intervention after 6-month delay (wait list control group)

INTERVENTIONS:
Behavioral: Many Men, Many Voices (3MV) — Small-group, 6-session HIV prevention intervention for Black MSM.
  Arms: Many Men, Many Voices (3MV) Intervention

SUMMARY:
The purpose of this program evaluation is to determine whether the "Many Men, Many Voices" HIV/STD prevention intervention is effective in reducing HIV sex risk behaviors and increasing HIV testing among African-American men who have sex with men (MSM), who may or may not self-identify as gay. The intent of this program is to support the evaluation of an existing intervention and provide feedback to the implementing organization for improved program effectiveness, not to conduct research.

DETAILED DESCRIPTION:
Black men who have sex with men (MSM) in the United States experience disproportionately high rates of HIV and other sexually transmitted infections (STIs); however, the number of evidence-based interventions for Black MSM is limited. This study evaluated the efficacy of Many Men, Many Voices (3MV), a small-group HIV/STI prevention intervention developed by Black MSM-serving community-based organizations and a university-based HIV/STI prevention and training program. The study sample included 338 Black MSM of HIV-negative or unknown HIV serostatus residing in New York city. Participants were randomly assigned to the 3MV intervention condition (n = 164) or wait-list comparison condition (n = 174). Relative to comparison participants, 3MV participants reported significantly greater reductions in any unprotected anal intercourse with casual male partners; a trend for consistent condom use during receptive anal intercourse with casual male partners; and significantly greater reductions in the number of male sex partners and greater increases in HIV testing. This study is the first randomized trial to demonstrate the efficacy of an HIV/STI prevention intervention for Black MSM.

ELIGIBILITY:
Inclusion Criteria:

* Black men who have sex with other men (i.e., self-identify as gay or bisexual or same gender-loving, or sexually active with other men and do not identify as gay or bisexual, or have sexual or emotional attraction to other men)
* 18 years of age or older
* Self-report their HIV serostatus as negative or unknown
* Willing to attend an intervention retreat (without their primary partner)
* Willing to discuss male-to-male sex
* Resident of the New York Metropolitan area and plan to reside in that area for at least 6 months
* Not previously participated in a Many Men, Many Voices intervention program

Exclusion Criteria:

* Individuals indicating an HIV positive serostatus
* Under 17 years of age
* Individuals not meeting the inclusion criteria specified above

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2005-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Painter, PhD, Study Director — Project Officer, Division of HIV/AIDS Prevention, NCHSTP, Centers for Disease Control and Prevention; Jeffrey H Herbst, PhD, Study Director — Project Officer, Division of HIV/AIDS Prevention, NCHSTP, Centers for Disease Control and Prevention
Locations (1):
- People of Color in Crisis, Inc., Brooklyn, New York, United States

REFERENCES:
- [Background] Coury-Doniger P, Wilton L, Herbst JH, Painter TM. HIV prevention interventions for black MSM. Am J Public Health. 2010 Feb;100(2):198. doi: 10.2105/AJPH.2009.182485. Epub 2009 Dec 17. No abstract available. PMID 20019294
- [Result] Wilton L, Herbst JH, Coury-Doniger P, Painter TM, English G, Alvarez ME, Scahill M, Roberson MA, Lucas B, Johnson WD, Carey JW. Efficacy of an HIV/STI prevention intervention for black men who have sex with men: findings from the Many Men, Many Voices (3MV) project. AIDS Behav. 2009 Jun;13(3):532-44. doi: 10.1007/s10461-009-9529-y. Epub 2009 Mar 9. PMID 19267264
- [Derived] Herbst JH, Painter TM, Tomlinson HL, Alvarez ME; Centers for Disease Control and Prevention (CDC). Evidence-based HIV/STD prevention intervention for black men who have sex with men. MMWR Suppl. 2014 Apr 18;63(1):21-7. PMID 24743663

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From August 2005 through November 2006, People of Color in Crisis Inc. recruited potential participants from venues throughout New York City.
Period: Overall Study
Arm/Group | Many Men, Many Voices (3MV) Intervention | Wait List Comparison
Started | 164 | 174
Complete 3-month Follow-up | 120 | 125
Completed 6-month Follow-up | 127 (7 participants who were lost to follow-up at 3-months were retained at 6-months) | 133 (8 participants who were lost to follow-up at 3-months were retained at 6-months)
Completed | 127 | 133
Not Completed | 37 | 41
Not completed — Lost to Follow-up | 37 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Many Men, Many Voices (3MV) Intervention | Wait List Comparison | Total
Number analyzed (Participants) | 164 | 174 | 338
Age Continuous [Mean (Standard Deviation); unit: years] | 29.5 (9.1) | 29.7 (9.5) | 29.6 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0.0
  Male | 164 | 174 | 338.0
Region of Enrollment [Number; unit: participants]
  United States | 164 | 174 | 338.0

OUTCOME MEASURES:

1. Primary Outcome: Any Unprotected Anal Intercourse (UAI) With Casual Partners
Description: Sexual activities with casual male partners in past 3 months (i.e., any unprotected insertive or receptive anal sex)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Number of episodes
Arm/Group | Many Men, Many Voices (3MV) Intervention | Wait List Comparison
Number analyzed (Participants) | 127 | 133
Number of episodes | 2.0 (5.6) | 6.2 (22.7)
Statistical Analysis 1: Comparison: Many Men, Many Voices (3MV) Intervention vs Wait List Comparison; Test type: Superiority or Other; p < 0.05, negative binomial regression; Rate Ratio = 0.58, 95% CI [0.33 to 1.01]

2. Primary Outcome: Number of Participants Reporting HIV Testing Behavior
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Many Men, Many Voices (3MV) Intervention | Wait List Comparison
Number analyzed (Participants) | 126 | 133
participants | 69 | 58
Statistical Analysis 1: Comparison: Many Men, Many Voices (3MV) Intervention vs Wait List Comparison; Test type: Superiority or Other; p < 0.05, generalized estimating equations; Tests intervention efficacy over all study periods (baseline, 3-months, and 6-months); Odds Ratio (OR) = 1.33, 95% CI [1.05 to 1.68]

3. Primary Outcome: Number of Participants Reporting Sexually Transmitted Disease (STD) Testing Behavior
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Many Men, Many Voices (3MV) Intervention | Wait List Comparison
Number analyzed (Participants) | 127 | 133
participants | 43 | 43
Statistical Analysis 1: Comparison: Many Men, Many Voices (3MV) Intervention vs Wait List Comparison; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Odds Ratio (OR) = 1.17, 95% CI [0.69 to 1.98]

4. Primary Outcome: Number of Episodes of Insertive Unprotected Anal Intercourse (UAI) With Casual Partners
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | Many Men, Many Voices (3MV) Intervention | Wait List Comparison
Number analyzed (Participants) | 127 | 133
number of episodes | 1.1 (3.4) | 4.5 (18.6)
Statistical Analysis 1: Comparison: Many Men, Many Voices (3MV) Intervention vs Wait List Comparison; Test type: Superiority or Other; p < 0.05, generalized estimating equations; Tests intervention efficacy over all study periods (baseline, 3-months, and 6-months); Rate Ratio = 0.49, 95% CI [0.28 to 0.87]

5. Primary Outcome: Number of Episodes of Receptive Unprotected Anal Intercourse (UAI) With Casual Partners
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | Many Men, Many Voices (3MV) Intervention | Wait List Comparison
Number analyzed (Participants) | 127 | 133
number of episodes | 0.9 (3.3) | 1.7 (6.8)
Statistical Analysis 1: Comparison: Many Men, Many Voices (3MV) Intervention vs Wait List Comparison; Test type: Superiority or Other; p < 0.05, generalized estimating equations; Tests intervention efficacy over all study periods (baseline, 3-months, and 6-months); Rate Ratio = 0.80, 95% CI [0.42 to 1.53]

ADVERSE EVENTS:
Arm/Group | Many Men, Many Voices (3MV) Intervention | Wait List Comparison
Serious Adverse Events (participants affected / at risk) | 0/164 | 0/174
Other Adverse Events (participants affected / at risk) | 0/164 | 0/174

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less